CLINICAL TRIAL: NCT06645821
Title: Open-label, Investigator-initiated, Single-site Proof of Concept Trial Evaluating EVO101 in Adult Subjects with Mild to Moderate Hidradenitis Suppurativa.
Brief Title: Participants with Mild to Moderate Hidradenitis Suppurativa Will Receive EVO101 a Topical Cream 0.1%
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Clinical Research, Inc. (Other)
Collaborators: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVO101-HS001
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: EVO101; Hidradenitis Suppurativa; topical cream; Acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label EVO101 topical cream 0.1% (Experimental): All eligible subjects will receive open label EVO101 topical cream 0.1%
  Interventions: Drug: EVO101

INTERVENTIONS:
Drug: EVO101 — EVO101 topical cream 0.1%

SUMMARY:
The goal of this clinical trial is to learn if drug EVO101 works to treat mild to moderate hidradenitis suppurativa in adults. The main questions it aims to answer are:

Does drug EVO101 lower the total number of lesion a participant has from the first visit to the last visit.

What medical problems do participants have when applying drug EVO101 Does a participant perceive a change in their hidradenitis suppurativa symptoms based on patient reported outcome questionnaires.

Participants will:

Apply EVO101 topical cream 0.1% topically Visit the clinic four times unless the first and second appointment have to be done separately then there will be five clinic visits and one phone call over a twelve week period.

Keep a dosing diary

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willingness to sign a written informed consent form (ICF) for the study.
2. Age ≥ 18 years at the time of signing the ICF (informed consent).
3. Diagnosis of hidradenitis suppurativa (HS) for at least 3 months prior to the screening visit.
4. Mild to moderate HS (hidradenitis suppurativa) at the Baseline Visit (using the HS-PGA/Hidradenitis Suppurativa Physician's Global Assessment scale ).
5. Total hidradenitis suppurativa lesion count (abscess, fistulas, nodules, papules, and/or pustules) of at least 5 at the baseline visit.
6. Agreement to NOT use topical and/or systemic antibiotics for treatment of HS (hidradenitis suppurativa) for the duration of the study.
7. Agreement to NOT use a diluted bleach bath or topical antiseptic washes containing chlorhexidine gluconate or benzoyl peroxide. Note: Over-the-counter non-medicated soap and water is allowed.
8. For women of childbearing potential: agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method during the treatment period and for at least 30 days after the last application of study drug.

   * A woman of childbearing potential is defined as a postmenarcheal female, who has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and/or uterus).
   * The following are highly effective contraceptive methods: combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) associated with inhibition of ovulation, progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, or sexual abstinence. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception. Females must agree not to donate ova during the study and for 30 days after the end of study visit.
9. Willing and able to comply with the study protocol and procedures.

Exclusion Criteria:

1. Very severe, severe, minimal, or clear hidradenitis suppurativa Hidradenitis Suppurativa Physician's Global Assessment scale (HS-PGA).
2. Women who are pregnant (or who are considering pregnancy) or breastfeeding.
3. Subject has uncontrolled, clinically significant comorbidities that make them unsuitable for the clinical trial in the opinion of the investigator.
4. Have undergone significant trauma or major surgery (per investigator's assessment) within 30 days preceding the screening visit.
5. History of clinically significant (per investigator's judgment) drug or alcohol abuse within 6 months preceding the screening visit.
6. Use of any of the following medications or treatments within the specified time periods prior to the baseline visit:

   1. < 12 weeks or 5 half-lives (whichever is longer)

      * Investigational or experimental treatments.
      * Immunomodulating biologic drugs
   2. < 4 weeks

      * Systemic JAK inhibitors.
      * Systemic immunosuppressive or immunomodulating small-molecule drugs (eg, corticosteroids [oral or intravenous], avacopan, IRAK4 inhibitors, methotrexate, cyclosporine, dapsone, azathioprine).
      * Surgical, laser, or any phototherapy intervention in areas with HS lesions
   3. < 2 weeks

      • Other systemic therapies for HS
      * Retinoids, antihyperglycemics, and antiandrogens, such as acitretin, isotretinoin, metformin, spironolactone, and finasteride) with potential therapeutic impact unless the subject is on a stable dose as defined by the investigator for at least 28 days. There should be no anticipated change of these medications while the subject is on the study.

        • Systemic anti-infectives for HS
      * Antibiotics, antivirals, antifungals
   4. <1 week

      * Oral or topical PDE4 inhibitor (e.g., apremilast, crisaborole)
      * Topical JAK inhibitor
      * Topical anti-infectives for HS lesions

        o Antibiotics, antivirals, antifungals
      * Topical products containing chlorhexidine gluconate, benzoyl peroxide, or topical diluted bleach bath to treat HS. Note: Non-medicated over-the-counter soap and water are not restricted.
      * Any topical drug applied onto HS lesions
      * Topical or intralesional corticosteroids o Note: Use of topical corticosteroids for dermatologic diseases other than HS (Hidradenitis Suppurativa)(e.g., atopic dermatitis, psoriasis) is allowed for areas not being treated for HS (Hidradenitis Suppurativa)as long as it is not within 10cm of the areas affected by HS (Hidradenitis Suppurativa).

   Inhaled corticosteroids are allowed.
7. Active participation in an experimental therapy study or who received experimental therapy within 30 days or 5 half-lives (whichever is longer) before Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The efficacy of EVO101 on hidradenitis suppurativa will be evaluated using two parameters: decrease in lesion count and change in patient reported outcomes (PRO) | 12 Weeks
  The change in the total HS lesion count will be assessed at Week 4, Week 8, and Week 12. The percent change from Baseline will be calculated.
The efficacy of EVO101 on hidradenitis suppurativa will be evaluated using two parameters: decrease in lesion count and change in patient reported outcomes (PRO) | 12 Weeks
  PRO's will be completed to evaluate whether the subjects perceive a change in their HS symptoms. PRO's will include the DLQI, NRS Scale of Pain, and Patient Impression of Severity. Efficacy will be calculated by the percent change in each PRO from Baseline at Week 4, Week 8, and Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Clinical Research, Inc., Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Lesion count and PRO data
Supporting Information: Study Protocol, CSR